CLINICAL TRIAL: NCT00868192
Title: Phase II Trial of Pemetrexed and Bevacizumab for Recurrent Ovarian and Primary Peritoneal Carcinoma
Brief Title: Trial of Pemetrexed and Bevacizumab for Recurrent Ovarian Primary Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0508 / 201102272
Record Dates: First submitted 2009-03-18; First posted 2009-03-24 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed and bevacizumab (Experimental): Pemetrexed 500 mg/m2 IV on Day 1 of each 21 day cycle
  Bevacizumab 15 mg/kg IV on Day 1 of each 21 day cycle
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed
  Other Names: Alimta
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine if the combination of bevacizumab and pemetrexed have an effect on recurrent ovarian and primary peritoneal carcinoma by looking at progression and survival at 6 months.

DETAILED DESCRIPTION:
Patients will be treated with pemetrexed 500 mg/m2 IV and Bevacizumab 15 mg/kg IV every 3 weeks.The patient is treated indefinitely until side effects are deemed severe by the investigator or until progression. Disease progression is measured every 6 weeks using RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian or primary peritoneal carcinoma. Histologic confirmation of the primary tumor is required. Patients with borderline tumors are not eligible.
* Patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in one dimension (longest dimension to be recorded). Each lesion must by > 20 mm when measured by conventional imaging techniques, including plain radiography, computed tomography and MRI or > 10 mm when measured by spiral CT.
* Patients must have at least one "target lesion" to assess response by RECIST criteria. Lesions within a previously irradiated field will be considered "non-target" lesions.
* Patients must have a GOG performance status of 0 or 1.
* Patients must have the ability to interrupt non-steroidal anti-inflammatory (NSAID) treatment 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed.
* Patients must have the ability to take folic acid, vitamin B12 and dexamethasone as described per protocol.
* Recovery from effects of recent surgery, radiotherapy or chemotherapy.
* Patients should be free of active infection requiring antibiotics.
* Any hormonal therapy directed at the tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy (HRT) is permitted.
* Any other prior therapy directed at the malignant tumor, including immunologic agents and cytotoxic agents, must be discontinued at least three weeks prior to registration.
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment.
* Patients must have had one prior regimen containing a taxane compound. Patient may have received first-line treatment either intravenously or intraperitoneally.
* Patients must NOT have received prior therapy with pemetrexed or bevacizumab.
* Patients may have received a total of < 2 prior cytotoxic chemotherapy regimens (adjuvant therapy plus one additional regimen). Consolidation or extended therapy as part of first line treatment will be considered as a single regimen.
* Bone marrow function: absolute neutrophil count (ANC) greater than or equal to 1,500/ul, equivalent to Common Toxicity Criteria (CTC) grade 1; Platelets greater than or equal to 100,000/ul.
* Creatinine clearance must be greater than 45 ml/min.
* Hepatic function: bilirubin less than or equal to 1.5 x ULN. AST and alkaline phosphatase less than or equal to 2.5 x ULN.
* Neurologic function: neuropathy (sensory and motor) less than or equal to CTC grade 1.
* Coagulation: prothrombin time (PT) such that the international normalized ratio (INR) is < 1.5 (INR may be between 2 and 3 if a patient is on stable dose of therapeutic warfarin) and a PTT < 1.2 times control.
* Patients must have signed informed consent.
* Patients must meet pre-entry requirements.
* Patients of childbearing potential must have a negative serum pregnancy test prior to study entry, be practicing an effective form of contraception, and cannot be lactating.
* Patients may have received prior radiotherapy (to less than 25% of bone marrow), but must start at a Level 1 dose reduction.

Exclusion Criteria:

* Patients with serious, non-healing wound, ulcer or bone fracture.
* Patients with clinically significant cardiovascular disease:
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* Unstable angina within 6 months prior to study enrollment.
* New York Heart Association (NYHA) grade II or greater congestive heart failure.
* Serious cardiac arrhythmia requiring medication.
* Grade II or greater peripheral vascular disease. Patients with claudication within 6 months.
* History of myocardial infarction within 6 months.
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
* Patients with the presence of ascites or other third space fluid which cannot be controlled by drainage.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of study or anticipation of need for major surgical procedure during the course of the study.
* Patients with history or evidence upon physical examination of central nervous system disease, including primary brain tumor, brain metastases, seizure not controlled with standard medical therapy, history of cerebrovascular accident (CVA, stroke), or transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
* Minor surgical procedures, other than central venous access placement, such as fine needle aspiration or core biopsy within 7 days prior to day 1 of study.
* Patients with proteinuria. At baseline patients will undergo a urine protein-creatinine ratio (UPCR) (Appendix IV). Patients with a UPCR > 1.0 at screening should be excluded. Urine dipstick for proteinuria may also be used. Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Patients whose circumstances do not permit completion of the study or the required follow-up.
* Patients who are pregnant or nursing.
* Patients under the age of 18.
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer within the last 5 years or whose previous cancer treatment contraindicates this protocol.
* Prior therapy with anti-angiogenic agents or pemetrexed.
* Patients with active infection requiring parenteral antibiotics.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months.
* Partial or complete small or large bowel obstruction demonstrated radiographically within 3 months prior to study.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study.
* Known hypersensitivity to any component of bevacizumab.
* Inability to comply with study and/or follow-up procedures.
* Life expectancy of less than 12 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Mutch, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. N Engl J Med. 1996 Jan 4;334(1):1-6. doi: 10.1056/NEJM199601043340101. PMID 7494563
- [Background] Alberts DS, Green S, Hannigan EV, O'Toole R, Stock-Novack D, Anderson P, Surwit EA, Malvlya VK, Nahhas WA, Jolles CJ. Improved therapeutic index of carboplatin plus cyclophosphamide versus cisplatin plus cyclophosphamide: final report by the Southwest Oncology Group of a phase III randomized trial in stages III and IV ovarian cancer. J Clin Oncol. 1992 May;10(5):706-17. doi: 10.1200/JCO.1992.10.5.706. PMID 1569443
- [Background] Ozols RF, Bundy BN, Greer BE, Fowler JM, Clarke-Pearson D, Burger RA, Mannel RS, DeGeest K, Hartenbach EM, Baergen R; Gynecologic Oncology Group. Phase III trial of carboplatin and paclitaxel compared with cisplatin and paclitaxel in patients with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2003 Sep 1;21(17):3194-200. doi: 10.1200/JCO.2003.02.153. Epub 2003 Jul 14. PMID 12860964
- [Background] Swenerton K, Jeffrey J, Stuart G, Roy M, Krepart G, Carmichael J, Drouin P, Stanimir R, O'Connell G, MacLean G, et al. Cisplatin-cyclophosphamide versus carboplatin-cyclophosphamide in advanced ovarian cancer: a randomized phase III study of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 1992 May;10(5):718-26. doi: 10.1200/JCO.1992.10.5.718. PMID 1569444
- [Background] Kosary CL. FIGO stage, histology, histologic grade, age and race as prognostic factors in determining survival for cancers of the female gynecological system: an analysis of 1973-87 SEER cases of cancers of the endometrium, cervix, ovary, vulva, and vagina. Semin Surg Oncol. 1994 Jan-Feb;10(1):31-46. doi: 10.1002/ssu.2980100107. PMID 8115784
- [Background] Folkman J. What is the evidence that tumors are angiogenesis dependent? J Natl Cancer Inst. 1990 Jan 3;82(1):4-6. doi: 10.1093/jnci/82.1.4. No abstract available. PMID 1688381
- [Background] Weidner N, Folkman J, Pozza F, Bevilacqua P, Allred EN, Moore DH, Meli S, Gasparini G. Tumor angiogenesis: a new significant and independent prognostic indicator in early-stage breast carcinoma. J Natl Cancer Inst. 1992 Dec 16;84(24):1875-87. doi: 10.1093/jnci/84.24.1875. PMID 1281237
- [Background] Weidner N, Semple JP, Welch WR, Folkman J. Tumor angiogenesis and metastasis--correlation in invasive breast carcinoma. N Engl J Med. 1991 Jan 3;324(1):1-8. doi: 10.1056/NEJM199101033240101. PMID 1701519
- [Background] Tammela T, Enholm B, Alitalo K, Paavonen K. The biology of vascular endothelial growth factors. Cardiovasc Res. 2005 Feb 15;65(3):550-63. doi: 10.1016/j.cardiores.2004.12.002. PMID 15664381
- [Background] Rosen LS. VEGF-targeted therapy: therapeutic potential and recent advances. Oncologist. 2005 Jun-Jul;10(6):382-91. doi: 10.1634/theoncologist.10-6-382. PMID 15967832
- [Background] Ferrara N, Kerbel RS. Angiogenesis as a therapeutic target. Nature. 2005 Dec 15;438(7070):967-74. doi: 10.1038/nature04483. PMID 16355214
- [Background] Zhang L, Yang N, Garcia JR, Mohamed A, Benencia F, Rubin SC, Allman D, Coukos G. Generation of a syngeneic mouse model to study the effects of vascular endothelial growth factor in ovarian carcinoma. Am J Pathol. 2002 Dec;161(6):2295-309. doi: 10.1016/s0002-9440(10)64505-1. PMID 12466143
- [Background] Goodheart MJ, Ritchie JM, Rose SL, Fruehauf JP, De Young BR, Buller RE. The relationship of molecular markers of p53 function and angiogenesis to prognosis of stage I epithelial ovarian cancer. Clin Cancer Res. 2005 May 15;11(10):3733-42. doi: 10.1158/1078-0432.CCR-04-0056. PMID 15897570
- [Background] Abulafia O, Ruiz JE, Holcomb K, Dimaio TM, Lee YC, Sherer DM. Angiogenesis in early-invasive and low-malignant-potential epithelial ovarian carcinoma. Obstet Gynecol. 2000 Apr;95(4):548-52. doi: 10.1016/s0029-7844(99)00608-0. PMID 10725487
- [Background] Alvarez AA, Krigman HR, Whitaker RS, Dodge RK, Rodriguez GC. The prognostic significance of angiogenesis in epithelial ovarian carcinoma. Clin Cancer Res. 1999 Mar;5(3):587-91. PMID 10100710
- [Background] Stone PJ, Goodheart MJ, Rose SL, Smith BJ, DeYoung BR, Buller RE. The influence of microvessel density on ovarian carcinogenesis. Gynecol Oncol. 2003 Sep;90(3):566-71. doi: 10.1016/s0090-8258(03)00367-6. PMID 13678725
- [Background] Bamberger ES, Perrett CW. Angiogenesis in epithelian ovarian cancer. Mol Pathol. 2002 Dec;55(6):348-59. doi: 10.1136/mp.55.6.348. PMID 12456770
- [Background] Gasparini G, Bonoldi E, Viale G, Verderio P, Boracchi P, Panizzoni GA, Radaelli U, Di Bacco A, Guglielmi RB, Bevilacqua P. Prognostic and predictive value of tumour angiogenesis in ovarian carcinomas. Int J Cancer. 1996 Jun 21;69(3):205-11. doi: 10.1002/(SICI)1097-0215(19960621)69:33.0.CO;2-6. PMID 8682589
- [Background] Hollingsworth HC, Kohn EC, Steinberg SM, Rothenberg ML, Merino MJ. Tumor angiogenesis in advanced stage ovarian carcinoma. Am J Pathol. 1995 Jul;147(1):33-41. PMID 7541612
- [Background] Orre M, Lotfi-Miri M, Mamers P, Rogers PA. Increased microvessel density in mucinous compared with malignant serous and benign tumours of the ovary. Br J Cancer. 1998 Jun;77(12):2204-9. doi: 10.1038/bjc.1998.367. PMID 9649134
- [Background] Obermair A, Wasicky R, Kaider A, Preyer O, Losch A, Leodolter S, Kolbl H. Prognostic significance of tumor angiogenesis in epithelial ovarian cancer. Cancer Lett. 1999 Apr 26;138(1-2):175-82. doi: 10.1016/s0304-3835(99)00005-1. PMID 10378790
- [Background] Sonmezer M, Gungor M, Ensari A, Ortac F. Prognostic significance of tumor angiogenesis in epithelial ovarian cancer: in association with transforming growth factor beta and vascular endothelial growth factor. Int J Gynecol Cancer. 2004 Jan-Feb;14(1):82-8. doi: 10.1111/j.1048-891x.2004.14202.x. PMID 14764033
- [Background] Paley PJ, Staskus KA, Gebhard K, Mohanraj D, Twiggs LB, Carson LF, Ramakrishnan S. Vascular endothelial growth factor expression in early stage ovarian carcinoma. Cancer. 1997 Jul 1;80(1):98-106. doi: 10.1002/(sici)1097-0142(19970701)80:13.0.co;2-a. PMID 9210714
- [Background] Shen GH, Ghazizadeh M, Kawanami O, Shimizu H, Jin E, Araki T, Sugisaki Y. Prognostic significance of vascular endothelial growth factor expression in human ovarian carcinoma. Br J Cancer. 2000 Jul;83(2):196-203. doi: 10.1054/bjoc.2000.1228. PMID 10901370
- [Background] Orre M, Rogers PA. VEGF, VEGFR-1, VEGFR-2, microvessel density and endothelial cell proliferation in tumours of the ovary. Int J Cancer. 1999 Apr 20;84(2):101-8. doi: 10.1002/(sici)1097-0215(19990420)84:23.0.co;2-5. PMID 10096239
- [Background] Hartenbach EM, Olson TA, Goswitz JJ, Mohanraj D, Twiggs LB, Carson LF, Ramakrishnan S. Vascular endothelial growth factor (VEGF) expression and survival in human epithelial ovarian carcinomas. Cancer Lett. 1997 Dec 23;121(2):169-75. doi: 10.1016/s0304-3835(97)00350-9. PMID 9570355
- [Background] Nakanishi Y, Kodama J, Yoshinouchi M, Tokumo K, Kamimura S, Okuda H, Kudo T. The expression of vascular endothelial growth factor and transforming growth factor-beta associates with angiogenesis in epithelial ovarian cancer. Int J Gynecol Pathol. 1997 Jul;16(3):256-62. doi: 10.1097/00004347-199707000-00011. PMID 9421092
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Yang JC, Haworth L, Sherry RM, Hwu P, Schwartzentruber DJ, Topalian SL, Steinberg SM, Chen HX, Rosenberg SA. A randomized trial of bevacizumab, an anti-vascular endothelial growth factor antibody, for metastatic renal cancer. N Engl J Med. 2003 Jul 31;349(5):427-34. doi: 10.1056/NEJMoa021491. PMID 12890841
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Burger RA, Sill MW, Monk BJ, Greer BE, Sorosky JI. Phase II trial of bevacizumab in persistent or recurrent epithelial ovarian cancer or primary peritoneal cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Nov 20;25(33):5165-71. doi: 10.1200/JCO.2007.11.5345. PMID 18024863
- [Background] Garcia AA, Hirte H, Fleming G, Yang D, Tsao-Wei DD, Roman L, Groshen S, Swenson S, Markland F, Gandara D, Scudder S, Morgan R, Chen H, Lenz HJ, Oza AM. Phase II clinical trial of bevacizumab and low-dose metronomic oral cyclophosphamide in recurrent ovarian cancer: a trial of the California, Chicago, and Princess Margaret Hospital phase II consortia. J Clin Oncol. 2008 Jan 1;26(1):76-82. doi: 10.1200/JCO.2007.12.1939. PMID 18165643
- [Background] Cannistra SA, Matulonis UA, Penson RT, Hambleton J, Dupont J, Mackey H, Douglas J, Burger RA, Armstrong D, Wenham R, McGuire W. Phase II study of bevacizumab in patients with platinum-resistant ovarian cancer or peritoneal serous cancer. J Clin Oncol. 2007 Nov 20;25(33):5180-6. doi: 10.1200/JCO.2007.12.0782. PMID 18024865
- [Background] Shih C, Chen VJ, Gossett LS, Gates SB, MacKellar WC, Habeck LL, Shackelford KA, Mendelsohn LG, Soose DJ, Patel VF, Andis SL, Bewley JR, Rayl EA, Moroson BA, Beardsley GP, Kohler W, Ratnam M, Schultz RM. LY231514, a pyrrolo[2,3-d]pyrimidine-based antifolate that inhibits multiple folate-requiring enzymes. Cancer Res. 1997 Mar 15;57(6):1116-23. PMID 9067281
- [Background] Alati T, Worzalla JF, Shih C, Bewley JR, Lewis S, Moran RG, Grindey GB. Augmentation of the therapeutic activity of lometrexol -(6-R)5,10-dideazatetrahydrofolate- by oral folic acid. Cancer Res. 1996 May 15;56(10):2331-5. PMID 8625328
- [Background] Ozcan C, Wong SJ, Hari P. Reversible posterior leukoencephalopathy syndrome and bevacizumab. N Engl J Med. 2006 Mar 2;354(9):980-2; discussion 980-2. No abstract available. PMID 16514715
- [Background] Glusker P, Recht L, Lane B. Reversible posterior leukoencephalopathy syndrome and bevacizumab. N Engl J Med. 2006 Mar 2;354(9):980-2; discussion 980-2. doi: 10.1056/NEJMc052954. No abstract available. PMID 16510760
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Jubb AM, Hurwitz HI, Bai W, Holmgren EB, Tobin P, Guerrero AS, Kabbinavar F, Holden SN, Novotny WF, Frantz GD, Hillan KJ, Koeppen H. Impact of vascular endothelial growth factor-A expression, thrombospondin-2 expression, and microvessel density on the treatment effect of bevacizumab in metastatic colorectal cancer. J Clin Oncol. 2006 Jan 10;24(2):217-27. doi: 10.1200/JCO.2005.01.5388. Epub 2005 Dec 19. PMID 16365183
- [Background] Bibikova M, Talantov D, Chudin E, Yeakley JM, Chen J, Doucet D, Wickham E, Atkins D, Barker D, Chee M, Wang Y, Fan JB. Quantitative gene expression profiling in formalin-fixed, paraffin-embedded tissues using universal bead arrays. Am J Pathol. 2004 Nov;165(5):1799-807. doi: 10.1016/S0002-9440(10)63435-9. PMID 15509548
- [Background] Bibikova M, Yeakley JM, Chudin E, Chen J, Wickham E, Wang-Rodriguez J, Fan JB. Gene expression profiles in formalin-fixed, paraffin-embedded tissues obtained with a novel assay for microarray analysis. Clin Chem. 2004 Dec;50(12):2384-6. doi: 10.1373/clinchem.2004.037432. No abstract available. PMID 15563488
- [Background] Fan JB, Yeakley JM, Bibikova M, Chudin E, Wickham E, Chen J, Doucet D, Rigault P, Zhang B, Shen R, McBride C, Li HR, Fu XD, Oliphant A, Barker DL, Chee MS. A versatile assay for high-throughput gene expression profiling on universal array matrices. Genome Res. 2004 May;14(5):878-85. doi: 10.1101/gr.2167504. PMID 15123585
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to participant enrollment on 05/28/2008 and closed to participant enrollment on 11/30/2010.
Period: Overall Study
Arm/Group | Pemetrexed and Bevacizumab
Started | 38
Completed | 34
Not Completed | 4
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 34
Stage [Number; unit: participants] — Staging
  * I:The cancer is only within the ovary(ies) or fallopian tube(s)
  * II:Cancer involves 1 or both ovaries or fallopian tube(s) with pelvic extension
  * III: Cancer involves 1 or both ovaries or fallopian tubes(s) with microscopically confirmed peritoneal metastases outside the pelvis and/or regional lymph node metastasis (also can be primary peritoneal cancer)
  * IV:Distant spreading (also can be primary peritoneal cancer)
  participants
    Stage I/II | 1
    Stage III | 27
    Stage IV | 6
Histology [Number; unit: participants]
  Serous | 24
  Endometriod | 2
  Mixed | 3
  Other | 5
Tumor grade [Number; unit: participants] — G1: The tissue is well-differentiated (contains many healthy-looking cells).
  G2: The tissue is moderately differentiated (more cells appear abnormal than healthy).
  G3:The tissue is poorly differentiated or undifferentiated (all or most cells appear abnormal).
  participants
    Grade 1 | 3
    Grade 2 | 1
    Grade 3 | 30
Pathologic diagnosis [Number; unit: participants]
  Ovarian | 27
  Fallopian tube | 1
  Primary peritoneal | 6
Gynecologic Oncology Group (GOG) Performance Status [Number; unit: participants] — GOG Performance Status
  * 0 = Fully active, unrestricted activities of daily living
  * 1 = Ambulatory, but restricted in strenuous activity
  participants
    0 | 22
    1 | 12
Prior number of chemotherapy regimens [Number; unit: participants]
  1 | 20
  2 | 14
Platinum-free interval [Number; unit: participants]
  <6 months | 12
  6-12 months | 11
  >12 months | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS = Period from study entry until disease progression, death, or date of last contact
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
percentage of participants | 56 [38 to 71]

2. Secondary Outcome: Distribution of Progression-free Survival (PFS)
Description: PFS = Period from study entry until disease progression, death, or date of last contact
Time Frame: Median follow-up was 25.7 months (range 3.0-47.2 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
months
  Platinum-free interval of <6 months | 6.7 [4.1 to 9.9]
  Platinum-free interval of 6-12 months | 4.7 [2.8 to 8.4]
  Platinum-free interval of >12 months | 16.8 [4.6 to 23.2]

3. Secondary Outcome: Distribution of Overall Survival (OS)
Description: OS = observed length of time from entry into the study to death or date of last contact
Time Frame: Median follow-up was 25.7 months (range 3.0-47.2 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
months
  Platinum-free interval of <6 months | 16.7 [7.5 to 33.4]
  Platinum-free interval of 6-12 months | 24.9 [6.2 to 28.6]
  Platinum-free interval of >12 months | 28.0 [6.0 to NA] — The upper bound of the 95% CI was not estimable for this group because of too few patients at risk.

4. Secondary Outcome: Toxicity Associated With Bevacizumab and Pemetrexed
Description: Detailed serious adverse events and other adverse events are shown in the adverse event module of the results.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
percentage of participants
  Grade 3/4 hematologic toxicity | 53
  Most common non-hematologic toxicity - fatigue | 94
  Grade 3 renal toxicity | 6
  Gastrointestinal toxicity | 91
  Subsequently developed hematologic malignancies | 6

5. Secondary Outcome: Frequency of Clinical Response
Description: As measured by RECIST criteria
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
participants
  Complete response | 0
  Partial response | 14
  Stable disease | 18
  Progressive disease | 2

6. Secondary Outcome: Gene Expression as Assessed by Illumina cDNA Mediated Annealing, Selection, Extension and Ligation (DASL) Microarray From Paraffin-embedded Tumor Specimens With Response to Pemetrexed and Bevacizumab
Time Frame: 6 months
Population: This outcome was not analyzed. Columbia University was to participate in this study but did not. They were to perform the correlative studies.
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Association Between Levels of Thymidylate Synthase, Dihydrofolate Reductase, and Glycinamide Ribonucleotide Formyl Transferase and Ovarian Response to Pemetrexed and Bevacizumab
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 0

8. Post Hoc Outcome: Overall Survival (OS)
Description: OS = observed length of time from entry into the study to death or date of last contact
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
percentage of participants | 79 [62 to 90]

9. Post Hoc Outcome: Progression-free Survival (PFS)
Description: PFS = Period from study entry until disease progression, death, or date of last contact
Time Frame: Median follow-up was 25.7 months (range 3.0-47.2 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
months | 7.9 [4.6 to 10.9]

10. Post Hoc Outcome: Overall Survival (OS)
Description: OS = observed length of time from entry into the study to death or date of last contact
Time Frame: Median follow-up was 25.7 months (range 3.0-47.2 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
months | 25.7 [15.4 to 29.8]

11. Post Hoc Outcome: Overall Response Rate
Description: Overall response rate = complete response + partial response
  Complete response = disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial response = at least a 30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be non unequivocal progression of non-target lesions and no new lesions.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 34
percentage of participants | 41 [25 to 59]

12. Post Hoc Outcome: CA-125 Response
Description: A CA-125 response was defined as at least a 50% reduction in CA-125 levels from a pretreatment sample following guidelines described by the Gynecological Cancer Intergroup.
Time Frame: 6 months
Population: 7 participants were not evauable by CA-125 criteria.
Measure: Number; unit: participants
Arm/Group | Pemetrexed and Bevacizumab
Number analyzed (Participants) | 27
participants
  50% CA-125 response | 17
  75% CA-125 response | 8
  No CA-125 response | 2

ADVERSE EVENTS:
Arm/Group | Pemetrexed and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 5/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed and Bevacizumab (N=34)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Small bowel obstruction (Gastrointestinal disorders) | 1
Thromobolic event (Vascular disorders) | 1
Septic embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed and Bevacizumab (N=34)
Anemia (Blood and lymphatic system disorders) | 28
Leukopenia (Investigations) | 28
Thrombocytopenia (Investigations) | 15
Neutropenia (Investigations) | 33
Allergy (Immune system disorders) | 11
Cardiovascular (Cardiac disorders) | 11
Impaired coagulation (Blood and lymphatic system disorders) | 6
Constitutional (General disorders) | 32
Rash (Skin and subcutaneous tissue disorders) | 23
Endocrine (Endocrine disorders) | 1
Gastrointestinal (Gastrointestinal disorders) | 27
Genitourinary (Renal and urinary disorders) | 6
Hemorrhage (General disorders) | 4
Infection/febrile neutropenia (Infections and infestations) | 14
Lymphatics (Blood and lymphatic system disorders) | 1
Metabolic (Metabolism and nutrition disorders) | 31
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2
Neurologic (Nervous system disorders) | 21
Ocular (Eye disorders) | 6
Pain (General disorders) | 29
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 16
Vascular (Vascular disorders) | 1
Auditory (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes